CLINICAL TRIAL: NCT06413654
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Clinical Study to Evaluate the Efficacy and Safety of B001 Injection in Aquaporin-4 Antibody Positive Patients With Neuromyelitis Optica Spectrum Disorder
Brief Title: A Clinical Study of B001 Injection in the Treatment of Neuromyelitis Optica Spectrum Disorders(NMOSD)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPH-B001-301
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B001 injection (Experimental)
  Interventions: Drug: B001
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: B001 — The subjects will receive IV dose of B001 on Day 1 and Day 15 of RCP
  Arms: B001 injection
Other: Placebo — The subjects will receive IV dose of placebo matched to B001 on Day 1 and Day 15 of the RCP
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of B001 injection in aquaporin-4 antibody positive patients with neuromyelitis optica spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed NMOSD patients;
2. Experienced at least 1 recurrence of NMOSD within 1 year or at least 2 recurrence within 2 years prior to screening;
3. The blood pregnancy tests were negative within 7 days before the first dose in fertile female subjects. The fertile subjects and the male subjects whose partner are fertile woman agree to use reliable contraception during the study period and within 6 months after the study drug discontinuation;
4. Volunteer to participate in clinical research; Fully understand and know the study and sign the informed consent; Willing to follow and able to complete all test procedures.

Exclusion Criteria:

1. Subjects with severe NMOSD were judged by the researcher to be unfit to participate in this study;
2. Subjects with chronic active immune system diseases undergoing systematic treatment;
3. Received anti-CD20 or other cell depletion therapy within 6 months before first dose;
4. Received the prescribed drug treatment at the prescribed time before first dose;
5. Subjects who have participated in any drug clinical trials within 28 days prior to the first dose;
6. Received hematopoietic stem cell transplantation、 lymphatic irradiation before first dose;
7. Pregnant or lactating women; Subjects with birth plans during the trial;
8. Subjects who had undergone major surgery within 2 months prior to screening or were scheduled to undergo major surgery during the trial;
9. Subjects with severe, progressive, or uncontrolled disease who have been assessed by the investigator to be at increased risk of participating in the study;
10. A history of gastrointestinal perforation and/or fistula within 6 months prior to screening;
11. Subjects who received a live or attenuated vaccine within 4 weeks prior to initial administration, or who plan to receive vaccination during the study period;
12. Subjects with severe or persistent infection currently or within the 1 months prior to screening;
13. Subjects with positive gamma interferon release test;
14. Subjects who currently have active hepatitis or have a history of severe liver disease;
15. Uncontrolled systemic disease, or any other reason the investigator deems inappropriate for inclusion;
16. Abnormal laboratory test results;
17. Subjects with a history of alcohol or drug abuse in the 6 months prior to screeing, or who are abusing;
18. Subjects with symptoms of severe mental illness who are clinically uncooperative;
19. Subjects who were unable to undergo magnetic resonance imaging during the study and who had other conditions that the investigator considered inappropriate to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to first NMOSD Attack During RCP | Approximately 48 weeks
  The NMOSD attack is defined as the presence of new or worsening symptom(s) related to NMOSD.

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) Score | Approximately 48 weeks
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS).
Change in Vision Acuity/ Low contrast visual acuity (VA/LCVA) | Approximately 48 weeks
  Change in VA/LCVA
Annualized relapse rate (ARR) | Approximately 3 years
  Annualized attack rate is defined as total number of attacks divided by total person years.
Change in Opticospinal Impairment Scale (OSIS) | Approximately 48 weeks
  Change in OSIS
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 3 years
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.

CONTACTS AND LOCATIONS:
Locations (51):
- China (51):
  - Beijing Anzhen Hospital，Capital Medical University, Beijing
  - Beijing Tiantan Hospital，Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - The First Medical Center of PLA General Hospital, Beijing
  - The Third Medical Center of PLA General Hospital, Beijing
  - Cangzhou Central Hospital, Cangzhou
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Huizhou First Hospital, Huizhou
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - First People's Hospital of Yunnan Province, Kunming
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanyang Central Hospital, Nanyang
  - Qilu Hospital of Shandong University (Qingdao), Qingdao
  - The First Hospital of China Medical University, Shenyang
  - Shenzhen Hospital of University of Hong Kong, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Taihe Hospital, Shiyan
  - First Hospital of Shanxi Medical University, Taiyuan
  - Shanxi Provincial People's Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Tongji Hospital, Wuhan
  - The Second Affiliated Hospital of the Chinese People's Liberation Army Air Force Medical University, Xi'an
  - Xi'an International Medical Center Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Xiamen University, Xiamen
  - Yan'an University Xianyang Hospital, Xianyang
  - Yantai Mountain Hospital in Yantai City, Yantai
  - The Central Hospital of Yongzhou, Yongzhou
  - Zaozhuang Municipal Hospital, Zaozhuang
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zigong First People's Hospital, Zigong